CLINICAL TRIAL: NCT06901622
Title: A Randomized Double-cohort Exploratory Clinical Study of Camrelizumab and Chemotherapy With or Without Anlotinib as First-line Treatment for Advanced Gallbladder Cancer and Extrahepatic Cholangiocarcinoma
Brief Title: Camrelizumab and Chemotherapy With or Without Anlotinib as First-line Treatment for Advanced Gallbladder Cancer and Extrahepatic Cholangiocarcinoma
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Hong Zong, Professor of Medicine, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTC-02
Record Dates: First submitted 2024-09-02; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-11

CONDITIONS: Gallbladder Cancer and Extrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Gallbladder Neoplasms; Cholangiocarcinoma | interventions — camrelizumab; anlotinib; 130-nm albumin-bound paclitaxel; S 1 (combination)

STUDY DESIGN:
Intervention Model Description: Randomized Double-cohort Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Camrelizumab, anlotinib, nab-paclitaxel, S-1
  Interventions: Drug: Camrelizumab, anlotinib, nab-paclitaxel, S-1
- Cohort 2 (Experimental): Camrelizumab, nab-paclitaxel, S-1
  Interventions: Drug: Camrelizumab, nab-paclitaxel, S-1

INTERVENTIONS:
Drug: Camrelizumab, anlotinib, nab-paclitaxel, S-1 — Initial treatment (4 cycles) Carrelizumab: 200 mg, day 1, iv, q3w. Anlotinib: 10 mg, taken orally once a day, day 1~14, q3w. For patients with intolerance, the dose can be reduced to 8 mg.
  Nab-paclitaxel: 200 mg/m^2, day 1, iv, q3w. (Patients with poor tolerance can be given on the 1st and 8th days, and the total dosage remains unchanged).
  S-1: 60 mg/day for body surface area <1.25 m^2; 80 mg/day for body surface area = 1.25~1.50 m^2; 100 mg/day for body surface area >1.50 m^2; 2 times a day, administered on days 1 to 14, 3 weeks as a treatment cycle.
  After 4 cycles of initial treatment, the feasibility of surgery was evaluated. Operable patients: radical surgical resection, followed by 4 cycles of S-1 combined with carrelizumab (up to 1 year). During postoperative treatment, the investigator determined whether local radiotherapy (CCRT) was required.
  Inoperable patients: carrelizumab + anlotinib + S-1 were treated until intolerance or disease progression.
  Arms: Cohort 1
Drug: Camrelizumab, nab-paclitaxel, S-1 — Initial treatment (4 cycles) Carrelizumab: 200 mg, day 1, intravenous drip, 3 weeks as a treatment cycle. Nab-paclitaxel: 200 mg/m^2, day 1, intravenous drip, 3 weeks as a treatment cycle. (Patients with poor tolerance can be given on the 1st and 8th days, and the total dosage remains unchanged).
  S-1: 60 mg/day for body surface area <1.25 m^2; 80 mg/day for body surface area = 1.25~1.50 m^2; 100 mg/day for body surface area >1.50 m^2; 2 times a day, administered on days 1 to 14, 3 weeks as a treatment cycle.
  After 4 cycles of initial treatment, the patient's surgical feasibility was evaluated.
  Operable patients: radical surgical resection, followed by S-1 (4 cycles) combined with carrelizumab treatment (up to 1 year). During postoperative treatment, the investigator determined whether local radiotherapy (CCRT) was required.
  Inoperable patients: carrelizumab + S-1 treatment until intolerance or disease progression.
  Arms: Cohort 2

SUMMARY:
To evaluate the efficacy and safety of camrelizumab and chemotherapy with or without anlotinib as first-line treatment for advanced gallbladder cancer and extrahepatic cholangiocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients voluntarily join this study, sign informed consent, and have good compliance;
* 2) Age: 18 to 75 years old, both men and women;
* 3) Unresectable locally advanced, unresectable recurrent or metastatic gallbladder cancer or extrahepatic bile duct cancer confirmed by pathological histology, and have not received systemic treatment; (according to RECIST version 1.1, at least one measurable lesion), tissue samples must be provided for biomarker analysis, and newly obtained tissues are preferred. Patients who cannot provide newly obtained tissues can provide 5-8 5um thick paraffin sections preserved in archives;
* 4) ECOG score: 0-1 points;
* 5) Estimated survival period ≥12 weeks;
* 6) Adequate organ function, and the following laboratory test values are required at the time of screening:
* ①Routine blood test standards must meet the following: Hemoglobin content (HB) ≥90g/L (no blood transfusion within 14 days); Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥80×10^9/L (no interleukin 11 or TPO used within 14 days); White blood cell count (WBC) ≥4.0×10^9/L (no granulocyte stimulating factor used within 14 days).
* ② Biochemical examinations must meet the following criteria: Serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); ALT and AST ≤2.5 ULN; Cr ≤1.5 ULN or creatinine clearance (CCr) ≥60 ml/min, (Cockcroft-Gault formula); Serum albumin ≥ 25 g/L (2.5 g/dL)
* 7) Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%);
* 8) Adequate coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
* 9)Females of childbearing potential must take effective contraceptive measures during the study and for at least 6 months after the last dose and chemotherapy. It is recommended to start taking contraceptive measures at least 3 months before the administration of the study drug; males who have not been sterilized must take effective contraceptive measures during the study and for at least 6 months after the last dose and chemotherapy. Contraceptive measures are recommended to be initiated at least 3 months before study drug administration.

Exclusion Criteria:

* 1) Patients who have received anlotinib hydrochloride treatment or any anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody treatment in the past;
* 2) Patients with a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* 3) Patients with active hepatitis B or C, active pulmonary tuberculosis;
* 4) Patients with liver metastasis burden accounting for more than 50% of the total liver volume;
* 5) CT showed clear ulcerative lesions or positive stool occult blood;
* 6) Self-reported history of abnormal bleeding (excluding epistaxis) one month before enrollment;
* 7) Patients who have received allogeneic bone marrow transplantation or organ transplantation in the past;
* 8) Congenital pulmonary fibrosis, drug-induced pneumonia, organizing pneumonia, or active pneumonia confirmed by CT;
* 9) Injection of live attenuated vaccine within 4 weeks before the start of the study, or expected to be injected with live attenuated vaccine during the trial or within 5 months after the end of the trial;
* 10) Systemic application of glucocorticoids or immunosuppressants within 2 weeks before the start of the trial (Note: inhaled glucocorticoids and mineralocorticoids are allowed);
* 11) Multiple factors that affect oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction, etc.);
* 12) ≥ NCI CTCAE grade 2 peripheral neuropathy;
* 13) Infection requiring antibiotics within 14 days before the start of the trial;
* 14) Patients with any severe and/or uncontrolled diseases, including: Patients with poor blood pressure control using antihypertensive drugs (systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥100 mmHg); patients with grade II or above myocardial ischemia or myocardial infarction, arrhythmia (including QT interval ≥480ms); patients with grade III-IV heart failure according to NYHA standards, or left ventricular ejection fraction (LVEF) <50% indicated by cardiac ultrasound examination; Active or uncontrolled severe infection; Liver disease such as cirrhosis, decompensated liver disease, chronic active hepatitis; Poorly controlled diabetes (fasting blood glucose (FBG) >10mmol/L); Urinalysis indicates urine protein ≥++, and confirms that the 24-hour urine protein quantification is >1.0 g;
* 15) Long-term unhealed wounds or fractures;
* 16) Abnormal coagulation function (INR>1.5 or APTT>1.5 × ULN), bleeding tendency or receiving thrombolytic or anticoagulant treatment. Known hereditary or acquired bleeding and thrombotic tendencies, such as hemophilia, coagulation disorder, thrombocytopenia, hypersplenism, etc. Those who have coughed up blood or coughed up half a teaspoon (2.5 ml) or more of blood per day within 2 months before entering the study. Those who have clinically significant bleeding symptoms or have a clear bleeding tendency within 3 months before entering the study, such as gastrointestinal bleeding, bleeding gastric ulcer, baseline stool occult blood ++ and above, or vasculitis, etc. Long-term anticoagulation treatment with warfarin or heparin is required, or long-term antiplatelet therapy is required (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day).
* 17) Major surgery (craniotomy, thoracotomy or laparotomy) within 4 weeks before the study, or major surgery is expected during the study treatment, or non-diagnostic surgery within 4 weeks before the start of the trial;
* 18) History of gastrointestinal perforation and/or fistula within 6 months before the treatment; or experience of arterial/venous thrombotic events, such as cerebrovascular accident (except stable cerebral infarction assessed by the investigator), deep vein thrombosis and pulmonary embolism;
* 19) Clinically significant pleural effusion, including any pleural effusion found during physical examination, pleural effusion that has been treated before or is still in need of treatment. Patients with only a small amount of pleural effusion and ascites but no symptoms can be selected if the investigators assess that they do not need treatment;
* 20) Patients with significant malnutrition;
* 21) Patients with a history of psychotropic drug abuse and inability to quit or with mental disorders;
* 22) Other histories of primary malignant tumors, except for the following: 1) Malignant tumors that have been completely relieved for at least 2 years before enrollment and do not require other treatment during the study; 2) Non-melanoma skin cancer or malignant lentigo that has been adequately treated and has no evidence of disease recurrence; 3) Carcinoma in situ that has been adequately treated and has no evidence of disease recurrence;
* 23) Pregnant or breastfeeding female patients;
* 24) Patients with serious concomitant diseases that, according to the investigators' judgment, endanger patient safety or affect the patient's completion of the study;
* 25)Participating in other trials within 30 days before the start of the trial, or planning to participate in other trials during the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate, ORR | Time Frame: about 2 years
  The RECIST1.1 standards were used to evaluate the efficacy of drugs.

SECONDARY OUTCOMES:
Disease Control Rate, DCR | Time Frame: about 2 years
Progression Free Survival, PFS | Time Frame: about 2 years
Event Free Survival, EFS | Time Frame: about 2 years
2-year Overall Surviva rate | Time Frame: about 2 years
Surgical resection rate | Time Frame: about 2 years
Incidence of Adverse events (AE) | Time Frame: about 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: Undecided